CLINICAL TRIAL: NCT07072364
Title: The Use of Video Aids Versus Usual Care for Reduction in Decisional Conflict in Fibroid Treatment
Brief Title: Videos to Aid Decision Making for Fibroid Treatment
Acronym: Fibroid AUB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: OptumRx (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBGYN-GYN-QI-1
Record Dates: First submitted 2025-06-02; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Uterine Bleeding; Decision Aid
Keywords: Abnormal uterine bleeding; Uterine fibroids; Decisional Conflict Scale; Educational videos
MeSH Terms: conditions — Uterine Hemorrhage; Metrorrhagia; Leiomyoma | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receive an educational video or not. The patients decisional conflict will be measured after receiving the intervention or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients will receive no additional education prior to their scheduled appointment to discuss uterine fibroids.
- Video (Experimental): Patients in this arm will receive a 5 minute educational video regarding symptoms, diagnosis and management options of uterine fibroids prior to their scheduled outpatient visit.
  Interventions: Behavioral: Video on uterine fibroids

INTERVENTIONS:
Behavioral: Video on uterine fibroids — Patients will be sent a link to a 5 minute video on uterine fibroids including their diagnosis, symptoms and treatment options prior to their scheduled appointment.
  Other Names: Video
  Arms: Video

SUMMARY:
Uterine fibroids are a common condition that can cause heavy and/or painful menstrual bleeding. There are many treatment options, but they vary in efficacy, side effects, short-term recovery and long-term implications for future fertility. Patients can have difficulty deciding between these options. In this study, the investigators will randomly assign patients seeking treatment for fibroids to receive an educational video on fibroids and their treatment, versus usual care (no video). The investigators will assess their decisional conflict with and without exposure to the video using a validated survey to see if exposure to the educational video helps them make decisions.

DETAILED DESCRIPTION:
Decisional conflict is defined as personal uncertainty regarding which course of action to take when choice among different options involves risk, regret, or challenge to personal life values. Some factors that influence decisional conflict are inadequate knowledge, unclear values, inadequate support, and the perception that an ineffective decision has been made. In this study, the investigators hope to target the factor of inadequate knowledge to see if an educational-style video can decrease decisional conflict in patients with fibroids. This will be completed via assessment using a validated decisional conflict scale score the DCS-10. DCS-10 scores range from 0 to 100 with a larger number indicating a higher level of decisional conflict. Scores above 37.5 are associated with decision delay. Through improving knowledge via an educational video about fibroids, the investigators wish to determine if decisional conflict can be minimized.

This will be a randomized, single-blinded trial. Patients in the intervention arm will be sent an educational video on fibroids prior to their visit to discuss fibroid treatment options. All patients will receive routine clinical care and counseling regarding treatment options at their visit. After the visit, patients will complete a DCS-10 survey. Survey instruments will be sent via text message using the Way to Health platform, timed to automatically send based on appointment date.

Pilot data shows an average post-visit DCS-10 score of 29 within this gynecologic population. With the recommended effect size of 0.4 in the literature on DCS-10, a sample size of 154 patients is needed. The investigators anticipate study recruitment will take approximately six months. Individual participation in the study will begin when patients are sent an invitation to participate soon after scheduling a visit to discuss fibroid treatment. It will end with a post-visit DCS-10 survey within one week of the visit. The survey will take approximately 5 minutes to complete and the video duration is 5 minutes, for a total of 10 minutes of participant time after enrollment. Based on the time between scheduling and completing this visit, the time between enrollment and final survey collection will be approximately 1-12 weeks. Chart review will occur to capture treatment decisions within 12 weeks of visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uterine fibroids
* Scheduled appointment to discuss management of fibroids in an outpatient clinical site associated with the Hospital of the University of Pennsylvania

Exclusion Criteria:

* Age <18 or >55
* Uterine or cervical cancer
* Cervical dysplasia grade 2-3 within the last 12 mo
* Pregnancy
* Menopause
* Decision made prior to the study intake to have a surgical procedure for treatment of fibroids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale | 1 weeks after appointment
  Patients complete a 10 question Decisional Conflict Scale 10 Item Version (DCS-10) via text message up to 1 week after their completed appointment. Each of the 10 questions asks patients on a 0-5 Likert scale. Higher scores indicate more decisional conflict. Minimum score of 0 = no decisional conflict. Maximum score of 40 = high decisional conflict.

SECONDARY OUTCOMES:
Treatment selected | 12 weeks post appointment
  Patients will be assigned one of four treatment options based on documentation from initial consultation or from chart review within 12 weeks after appointment completion.
  1. Expectant management, defined as no medical or surgical intervention
  2. Medical management, defined as acceptance of prescribed medications such as oral contraceptive pills, GnRH modifiers (oral or injected), Injectable medications (such as Depo-Provera), Intrauterine devices.
  3. Surgical management, defined as myomectomy or hysterectomy.
  4. Other procedural management, defined as uterine artery embolization or high intensity focused ultrasound.
Time to treatment | 12 weeks post appointment
  Patients time to selected treatment will be determined based on documentation within the medical chart with regards to acceptance of treatment.
  1. Expectant management group, based on documentation within the medical record from initial visit.
  2. Medical management group, based on the date of prescription of medication or date of documented decision for intrauterine device placement.
  3. Surgical management group, based on the date of decision for surgical intervention as confirmed by scheduled procedure in chart.
  4. Other procedural management group, based on the date of decision for management as confirmed by scheduled appointment in chart.
Length of visit | Baseline
  Length of visit will be collected for all patients at baseline visit. This information is accessible by reviewing documented billing codes and documentation within the note from providers. Specifically for telehealth visits total minutes are available for all patients. If total time is not documented, pts will be assigned by level of visit billed to low end of the billable minutes.
  Level 2 10-19 min (assigned time would be 10 min) Level 3 20-29 min (assigned time would be 20 min) Level 4 30-39 min (assigned time would be 30 min) Level 5 40-54 min (assigned time would be 50 min)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Dokras, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Privacy concerns, not applicable to primary outcome.